CLINICAL TRIAL: NCT02322476
Title: Herpes Simplex Reactivation in Adult Critical Care Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Søren Aalbæk Madsen, MD, Rigshospitalet, Denmark
Other Study IDs: HSV-ITA-RH
Record Dates: First submitted 2014-11-19; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Herpes Simplex I; Herpes Simplex II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood tracheal secretions
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention will be performed — No intervention will be performed

SUMMARY:
Welcome or not Herpes Simplex virus (HSV) is an ever present guest in the intensive care unit (ICU). Several studies have documented a high frequency of HSV reactivation in critically ill patients despite that clinical impact remains unknown.

DETAILED DESCRIPTION:
Normally primary HSV infection is asymptomatic but can under certain circumstances cause manifestations such as encephalitis and bronchopneumonitis. Bruynseels showed that HSV was detectable in the throat of two percent of healthy volunteers and three percent of patients not admitted to the ICU, this provides a broad "recruitment-base" for either latent or lytic HSV infection in the ICU. Viral dissemination to the bloodstream is seen in neonates , immunocompromised patients, but also in patients with primary herpetic gingivostomatitis. Patients testing polymerase chain reaction (PCR) positive for herpes simplex DNA in blood, have a higher rate of systemic symptoms than those testing PCR negative for herpes simplex. Additionally it is known that HSV suppression in HIV patients has beneficial effects. PCR, now being available for more than a decade, has been shown to provide a more sensitive method for the detection of HSV than culture, but viral detection does not per se translate to viral disease thus the impact of disseminated HSV infection in ICU patients remains unclear.

The investigators would like to investigate the incidence of HSV reactivation in blood and tracheal secretions critically ill patients and its impact on clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU
* Expected length of stay (LOS) >72 hours
* Intubated <24 hours prior to inclusion
* Informed consent by patient, relative or guardian

Exclusion Criteria:

* Ongoing antiviral treatment/prophylaxis
* Expected LOS <72 hours
* Intubation >24 hours prior to inclusion
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-02 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of HSV reactivation | Approximately 16 days
  Participants will be followed for the duration of the hospital stay with sampling of blood or tracheal secretions every 4 days until end of the viral reactivation period

SECONDARY OUTCOMES:
Duration of mechanical ventilation | Approximately 16 days
  Participants will be followed for the duration of the hospital stay with sampling of blood or tracheal secretions every 4 days until end of the viral reactivation period
ICU length of stay | Approximately 16 days
  Participants will be followed for the duration of the hospital stay with sampling of blood or tracheal secretions every 4 days until end of the viral reactivation period
30/90 day mortality | 30/90 days